CLINICAL TRIAL: NCT01781884
Title: Effects Of Gamma Aminobutyric Acid On The Progression Of New Onset Juvenile
Brief Title: Effects Of Gamma Aminobutyric Acid On The Progression Of New Onset Juvenile Type 1 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Zhaoyun Zhang, clinical professor, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-024
Record Dates: First submitted 2013-01-12; First posted 2013-02-01 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — gamma-Aminobutyric Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Gamma Aminobutyric Acid (GABA) (Active Comparator): GABA will be given 50mg/kg/Day, thrice daily for 52 weeks
  Interventions: Drug: Gamma Aminobutyric Acid (GABA)
- Gamma Aminobutyric Acid GABA) (Active Comparator): GABA will be given 100mg/kg/Day, thrice daily for 52 weeks.
  Interventions: Drug: Gamma Aminobutyric Acid (GABA)
- placebo (Placebo Comparator): placebo will be given thrice daily for 52 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gamma Aminobutyric Acid (GABA) — two dosages will be used in this study. GABA: 50mg/kg/day and 100mg/kg/day
  Other Names: Gamma Aminobutyric Acid
  Arms: Gamma Aminobutyric Acid (GABA); Gamma Aminobutyric Acid GABA)
Drug: Placebo
  Arms: placebo

SUMMARY:
This study is a multicenter, randomized, double-masked, placebo-controlled clinical study. All groups will receive standard intensive diabetes treatment with insulin and life style management. 60 subjects will be randomly assigned in a 1:1:1 ratio to receive placebo or different dosage of GABA.

GABA is an amino acid produced from glutamate by glutamic acid decarboxylase. It was approved for the treatment of hepatic coma, fibromyalgia, ataxia in China and is widely used as supplement for the treatment of epilepsy, insomnia, stress and tobacco dependence. It has been recently shown that GABA can prevent and reverse the development of diabetes in type 1 mice models. Participants will receive placebo or GABA for 52 weeks.

The study will consist of 4 weeks screening period, 2 weeks run-in period, 52 weeks treatment period and 4 weeks follow-up period. Enrollment is expected to occur over 2 years.

To assess the efficacy and safety of GABA for the treatment of juvenile type 1 diabetes in new onset subjects.

DETAILED DESCRIPTION:
Primary Outcome:

The primary statistical hypothesis to be assessed in this study is whether the mean C-peptide value for study subjects receiving GABA differs significantly from the mean value for placebo subjects assessed at follow-up.

Secondary Outcome:

The study will examine the HbA1C and the daily dosage of insulin (units/kg).

Exploratory Endpoint:

The study will assess the effects of treatment on inflammatory markers and immunological outcomes.

Major Inclusion Criteria:

Type 1 diabetes within past 6 months Age 5-21 years* At least one diabetes associated autoantibody

ELIGIBILITY:
Inclusion Criteria:

1. Be between the ages of 5 and 21 years*
2. Be within 6-months of diagnosis of type 1 diabetes based on American Diabetes Association (ADA) criteria
3. Must have stimulated C-peptide levels ≥0.2 pmol/ml measured during a mixed meal tolerance test (MMTT) conducted at least 21 days from diagnosis of diabetes and within one month of randomization
4. Presence of at least one diabetes-related autoantibody
5. Must be willing to comply with intensive diabetes management and monitor glucose with glucometer.
6. If participant is female with reproductive potential, she must be willing to avoid pregnancy during the whole study period and have a negative pregnancy test
7. Parents and participants must sign the informed consent

Exclusion Criteria:

1. Be currently pregnant or lactating or anticipate getting pregnant during the study period.
2. Type 2 diabetes and other specific types of diabetes.
3. Require use of systemic immunosuppressant, steroids or other medications that can affect glucose metabolism.
4. Have a history of malignancies
5. Be currently using non-insulin pharmaceuticals to affect glycemic control
6. Have any acute or chronic complicating medical issues or abnormal clinical laboratory results that interfere with study conduct or cause increased risk.
7. Have a history of epilepsy, significant head trauma or cerebrovascular accident or clinical features of continuous motor unit activity in proximal muscles
8. Inability or unwillingness to comply with the provisions of this protocol
9. Have an active infection or positive PPD test result.
10. Have serologic evidence of current or past HIV, Hep B, or Hep C infection.
11. Be with acute complications of diabetes (diabetic ketoacidosis, nonketotic hypersmolar coma, diabetic lactic acidosis)
12. Have a history of chronic renal failure, serum creatinine higher than 177umol/L
13. Have a history of impaired liver function, ALT or AST level elevated more than (or equal to) 2.5 times of upper limmit normal.

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
C-peptide value | baseline and up to 52 weeks
  The primary statistical hypothesis to be assessed in this study is whether the mean C-peptide value for study subjects receiving GABA differs significantly from the mean value for placebo subjects assessed at follow-up.

SECONDARY OUTCOMES:
HbA1C level | baseline and up to 52 weeks
  The study will examine the HbA1C level every 3 months from baseline and up to 52 weeks.

OTHER OUTCOMES:
Daily dosage of insulin (units/kg). | baseline and up to 52 weeks
  The study will assess the daily dosage of insulin (units/kg).

CONTACTS AND LOCATIONS:
Overall Officials: Yiming Li, Doctor, Principal Investigator — Huashan Hospital; Qinghua Wang, Doctor, Principal Investigator — St Michale's Hospital, University of Toronto
Locations (1):
- Department of Endocrinology and Metabolism，Huashan hospital, Shanghai, Shanghai Municipality, China